CLINICAL TRIAL: NCT05207657
Title: Phase I/II, Non-randomised, Single-centre, Open-label Study of pCHIM-p47 (Lentiviral Vector Transduced CD34+ Cells) in Patients With p47 Autosomal Recessive Chronic Granulomatous Disease
Brief Title: Lentiviral Gene Therapy for p47 AR-CGD
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Great Ormond Street Hospital for Children NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19IC05
Record Dates: First submitted 2021-06-24; First posted 2022-01-26 (Actual); Last update posted 2023-05-16 (Actual); Status verified 2023-03

CONDITIONS: P47-Phox, Deficiency of
MeSH Terms: conditions — Granulomatous Disease, Chronic, Autosomal Recessive, Cytochrome B-Positive, Type I

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lentiviral vector transduced CD34+ cells (Experimental): The investigational product is patient-specific and corresponds to cryopreserved autologous CD34+ cells transduced ex vivo with the pCHIM-p47 vector containing the human p47phox (NCF1) gene in final formulation and container closure system, ready for intended medical use. The starting materials used for the production of the investigational product consist of the viral vector and the patient's CD34+ cells.
  Interventions: Drug: Lentiviral vector transduced CD34+ cells

INTERVENTIONS:
Drug: Lentiviral vector transduced CD34+ cells — Gene therapy for p47 AR-CGD will be performed by introduction a normal copy of the NCF-1 gene into the blood forming stem cells (CD34+ cells) of the patient's bone marrow by using a type of gene delivery system (in this trial called a lentiviral vector). The gene corrected cells are then transplanted back into the patient
  Other Names: p47LV transduced autologous CD34+ cells

SUMMARY:
Chronic Granulomatous Disease (CGD) is a rare inherited disorder in which patients suffer from severe infection and inflammation. The first indications of disease usually appear in early childhood. The basic defect has been found to be lie in specialised white blood cells called phagocytic cells, which are responsible for engulfing and destroying germs. In CGD, there is a defect in an enzyme (known as the NADPH-oxidase) that is responsible for generating bleach like substances that are important for killing some important germs. In one form of the disease known as p47 AR-CGD (which accounts for 30% of patients), there are defined mistakes in a gene called NCF1. This gene is needed to form a key component of NADPH-oxidase.

In many cases, patients can be protected from infection by constant intake of antibiotics. However, in others potentially life-threatening infections break through. In some cases patients also develop serious inflammation requiring high doses of drugs such as steroids. CGD can be cured by bone marrow transplant and the best results are available when a matched sibling donor is available. Transplant from unmatched donors have a much worse outcome and as a result alternative treatments for patients without a matched donor are highly desirable.

Gene therapy of p47 AR-CGD is performed by introducing a normal copy of the human NCF-1 gene into the blood forming stem cells in the patients' bone marrow by using a gene carrier (in this study called a lentiviral vector). After treatment of the bone marrow cells in a specialised laboratory they are given back to the patient and will grow into functional phagocytic cells. There have been no previous clinical trials for patients with p47 AR-CGD however there have been previous gene therapy clinical trials conducted in the UK for patients with the most common form of CGD, known as X-CGD.

ELIGIBILITY:
Inclusion Criteria:

1. p47 AR-CGD patients > 23 months of age
2. Molecular diagnosis confirmed by Deoxyribonucleic acid (DNA) sequencing and supported by laboratory evidence for absent or reduction > 95% of the biochemical activity of the NAHPD-oxidase
3. At least one prior, ongoing or refractory severe infection and/or inflammatory complications requiring hospitalisation despite conventional therapy
4. No 10/10 human leukocyte antigen (HLA)-matched donor available after initial search of National Marrow Donor Program (NMDP) registries performed within the last year
5. No co-infection with Human Immunodeficiency Virus (HIV) or hepatitis B virus (HBsAg positive) or hepatitis C virus (HCV ribonucleic acid (RNA) positive), Cytomegalovirus (CMV), adenovirus, parvovirus B 19 or toxoplasmosis
6. Written informed consent for adult patient
7. Parental/guardian and, where appropriate, child's signed consent/assent

Exclusion Criteria:

1. Age ≤ 23 months or > 35 kg body weight
2. 10/10 HLA identical (A,B,C,DR,DQ) family or unrelated adult donor unless there is deemed to be an unacceptable risk associated with an allogeneic procedure
3. Contraindication for leukapheresis (Haemoglobin <8g/dl, cardiovascular instability, severe coagulopathy)
4. Appropriate organ function as outlined below must be observed within 8 weeks of entering this trial.

   a) Haematologic i) Anaemia (hemoglobin < 8 g/dl). ii) Neutropenia (absolute granulocyte count <1,000/mm3 iii) Thrombocytopenia (platelet count < 150,000/mm3). iv) Prothrombin Time (PT) or Partial thromboplastin time (PTT) > 2 X the upper limits of normal (ULN) (patients with a correctable deficiency controlled on medication will not be excluded).

   v) Cytogenetic abnormalities known to be associated with haematopoietic defect on peripheral blood or bone marrow.

   b) Infectious i) Evidence of infection with HIV-1 and -2, hepatitis B, Hepatitis C, adenovirus, parvovirus B 19 or toxoplasmosis within 8 weeks prior to mobilisation/pheresis or bone marrow harvest. CMV infection is allowable as long as the infection is under control.

   c) Pulmonary i) Resting O2 saturation by pulse oximetry < 90% on room air. d) Cardiac i) Abnormal electrocardiogram (ECG) indicating cardiac pathology. ii) Uncorrected congenital cardiac malformation with clinical symptomatology. iii) Active cardiac disease, including clinical evidence of congestive heart failure, cyanosis, iv) Hypotension. v) Poor cardiac function as evidenced by Left Ventricular Ejection Fraction (LVEF) < 40% on echocardiogram.

   e) Neurologic i) Significant neurologic abnormality by examination. ii) Uncontrolled seizure disorder. f) Renal i) Renal insufficiency: serum creatinine greater than or equal to 1.5 mg/dl, or greater than or equal to 3+ proteinuria ii) Abnormal serum sodium, potassium, calcium, magnesium at grade III or IV according to the Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 g) Hepatic/GI: i) Serum transaminases > 5X the upper limit of normal (ULN). ii) Serum Bilirubin > 2X ULN. iii) Serum Glucose > 1.5x ULN. h) Oncologic i) Evidence of active malignant disease
5. General

   1. Expected survival < 6 months.
   2. Major congenital anomaly.
   3. Ineligible for autologous Haematopoietic Stem Cell Transplant (HSCT) by the criteria at the clinical site.
   4. Contraindication for administration of conditioning medication
   5. Known sensitivity to Busulfan
6. Administration of gamma-interferon within 30 days before the infusion of transduced, autologous CD34+ cells
7. Participation in another experimental therapeutic protocol within 6 months prior to baseline and during the study period
8. Any other condition that, in the opinion of the Investigator, may compromise the safety or compliance of the patient or would preclude the patient from successful study completion
9. Patient/Parent/Guardian unable or unwilling to comply with the protocol requirements.

Min Age: 23 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2023-03-20 (Actual); Primary Completion 2029-04-01 (Estimated); Study Completion 2029-04-01 (Estimated)

PRIMARY OUTCOMES:
To evaluate the safety of p47 LV transduced autologous CD34+ cells treatment in p47 AR-CGD patients. | 6 months to 1 year
  The safety will be measure by:
  * Safety of the gene therapy procedure will be assessed through evaluation of adverse reactions after infusion and adverse reactions observed by the investigator or reported by the patient/parent/guardian during the study period.
  * As part of the overall safety evaluation, analysis of the lentivirus integration sites will be performed in different cell subpopulations and to investigate specific clonal expansions. Quantification of transgene copy numbers is determined on sorted cell populations by ddPCR methodology.
To evaluate the efficacy of p47 LV transduced autologous CD34+ cells treatment in p47 AR-CGD patients. | 6 months to 1 year
  Failure of gene therapy is defined by the absence of the NCF1 functioning granulocytes assessed by a DHR test (< 5% of expressing cells) 12 months after the procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Claire Booth, Principal Investigator — UCL Great Ormond Street Institute of Child Health
Locations (1):
- Great Ormond Street Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No